CLINICAL TRIAL: NCT01628380
Title: Stage IIIC Unresectable Epithelial Ovarian/Tubal Cancer With Partial or Complete Response After 1st Line Neoadjuvant Chemotherapy (3 Cycles CBDCA+Paclitaxel): a Phase 3 Prospective Randomized Study Comparing Cytoreductive Surgery + Hyperthermic Intraperitoneal Chemotherapy (CDDP+Paclitaxel) + 3 Cycles CBDCA+Paclitaxel vs Cytoreductive Surgery Alone + 3 Cycles CBDCA+Paclitaxel.
Brief Title: Phase 3 Trial Evaluating Hyperthermic Intraperitoneal Chemotherapy in Upfront Treatment of Stage IIIC Epithelial Ovarian Cancer
Acronym: CHORINE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: A.O. Ospedale Papa Giovanni XXIII (Other)
Collaborators: Clinical Organization for Strategies & Solutions (CLIOSS), former Nerviano Medical Sciences (http://www.nervianoms.com/en/) (Unknown); Onlus Cancro Primo Aiuto (http://www.cpaonlus.it/) (Unknown)
Responsible Party: Principal Investigator, Luca Ansaloni MD, MD, A.O. Ospedale Papa Giovanni XXIII
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHORINE 2012-002616-22
Record Dates: First submitted 2012-06-22; First posted 2012-06-26 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Ovarian Neoplasms
Keywords: HIPEC; Ovarian Cancer; Cytoreductive Surgery
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Cytoreduction Surgical Procedures; Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CRS + HIPEC (Active Comparator): Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy with CDDP+Paclitaxel
  Interventions: Procedure: Cytoreductive Surgery and HIPEC
- CRS alone (Active Comparator): Cytoreductive Surgery alone
  Interventions: Procedure: CRS alone

INTERVENTIONS:
Procedure: Cytoreductive Surgery and HIPEC — CRS: radical surgery, associated to any surgical procedure needed to obtain a zero or ≤ 0.25cm residual tumor (peritonectomy, bowel resection, diaphragmatic stripping, gastric resection, etc.).
  HIPEC: Cisplatin (CDDP) (100 mg/m2 of body surface area) + Paclitaxel (175mg/m2 of body surface area). Closed/open technique, as preferred. Duration: 90 minutes. Mean Intra-abdominal Temperature: 42°C.
  Arms: CRS + HIPEC
Procedure: CRS alone — CRS: radical surgery, associated to any surgical procedure needed to obtain a zero or ≤ 0.25cm residual tumor (peritonectomy, bowel resection, diaphragmatic stripping, gastric resection, etc.)
  Arms: CRS alone

SUMMARY:
Aim of the Study is to compare two-years disease-free survival of Cytoreductive Surgery (CRS) and Hyperthermic IntraPEritoneal Chemotherapy (HIPEC, CDDP+Paclitaxel) vs CRS alone in Stage IIIC unresectable epithelial tubal/ovarian cancer with partial or complete response after 3 cycles of 1st line chemotherapy (CBDCA +Paclitaxel).

DETAILED DESCRIPTION:
Eligible: Female adult women (18 to 70 years old) patients, with epithelial ovarian/tubal (FIGO stage IIIC) with a Fagotti modified Laparoscopic Scoring System ≥ 4 who will show a complete or partial clinical response(RECIST 1.1) after 3 cycles of neoadjuvant chemotherapy (Carboplatin+Paclitaxel).

Duration of recruitment: 2 years. Sample size has been calculated to reach a confidence level of 95% with a power of 80%, considering a 45% and 75% disease-free survival at 2 years in CRS and CRS+HIPEC group respectively.

Sample size will be 47 patients for each group. After CRS, only patients with adequate cytoreduction (CC 0-1, residual tumor ≤ 2.5mm) will be randomized. Patients with suboptimal cytoreduction (CC 2-3, residual tumor > 2.5mm) are not suitable for randomization.

The drug schedule elected in the current study is Cisplatin (CDDP) (100 mg/m2 of body surface area) + Paclitaxel (175mg/m2 of body surface area).

Closed/open technique, as preferred. Duration: 90 minutes. Mean Intra-abdominal Temperature: 42°C. Primary Endpoint: 2-years disease-free survival.

Secondary Endpoints:

1-year, 3- and 5-years disease-free survival;

1 month, 1-year, 3- and 5-years overall survival; toxicity induced by HIPEC using the NCI CTC criteria; one month and six months morbidity; duration of operation; return of bowel function; length of hospital stay; return to normal activity; six months and one year QOL, using the SF-36 v1.0; percentage of patients in both arms completing the scheduled postoperative chemotherapy; Subgroup analysis: PCI ≤ 15; pts. ≤ 40yrs.

Main topics of this Study:

Focused only on upfront treatment of primary disease. Select platinum-sensible patients (responders to platinum-based neoadjuvant chemotherapy).

Take advantage of NACT to maximize chances for cytoreduction. Standardized strategy for CRS: radical surgery, associated to any surgical procedure needed to obtain a zero or ≤ 0.25cm residual tumor (peritonectomy, bowel resection, diaphragmatic stripping, gastric resection, etc.). Pelvic and peri-aortic lymphadenectomy is not chosen as standard procedure, but should warrant adequate staging.

Compare only the effect of HIPEC.

ELIGIBILITY:
Inclusion Criteria:

* Female adult women (18 to 70 years old) patients, with EOC (FIGO stage IIIc) with a Fagotti modified Laparoscopic Scoring System ≥ 4 who will show a complete clinical response (cCR) or partial clinical response (cPR) after 3 cycles (Carboplatin+Paclitaxel) of neoadjuvant chemotherapy;
* performance status (ECOG) 0, 1 or 2;
* signed informed consent.

Exclusion Criteria:

* refusing to sign an informed consent;
* age > 70 years and age <18 years;
* BMI > 35;
* impossibility of an adequate follow-up;
* presence of other active neoplasms;
* active infection or other concurrent medical condition that could interfere in the ability of patients to receive the proposed treatment according to protocol;
* extraabdominal metastases (Stage IV) ;
* performance status (ECOG)>2;
* complete bowel obstruction;
* Abnormal bone marrow indices or renal and liver function;
* ASA IV or V.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2012-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 2 years

SECONDARY OUTCOMES:
postoperative morbidity and mortality | 1 and 6 months
Time to Chemotherapy | 3 months
  percentage of patients in both arms completing the scheduled postoperative chemotherapy and time elapsed to start postoperative chemotherapy
Overall Survival | 1, 3 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Luca Ansaloni, MD, Principal Investigator — A.O. Ospedale Papa Giovanni XXIII
Locations (5):
- Jena University Hospital, Jena, Germany
- Italy (4):
  - A.O. Papa Giovanni XXIII (former Ospedali Riuniti), Bergamo, Bg
  - A.O. Universitaria Policlinico S.Orsola-Malpighi Di Bologna - Bologna (Bo), Bologna, Bo
  - A.O. Universitaria Di Parma - Parma (Pr) Oncologia Chirurgica, Parma, Pr
  - POLICLINICO UNIVERSITARIO GEMELLI DI ROMA - ROMA (RM) GINECOLOGIA E OSTETRICIA Dipartimento per la Tutela della Salute della Donna e della Vita Nascente, Roma, Roma

REFERENCES:
- [Background] Ansaloni L, De Iaco P, Frigerio L. Re: "cytoreductive surgery and hyperthermic intraperitoneal chemotherapy as upfront therapy for advanced epithelial ovarian cancer: multi-institutional phase II trial." - Proposal of a clinical trial of cytoreductive surgery and hyperthermic intraperitoneal chemotherapy in advanced ovarian cancer, the CHORINE study. Gynecol Oncol. 2012 Apr;125(1):279-81. doi: 10.1016/j.ygyno.2012.01.001. Epub 2012 Jan 9. No abstract available. PMID 22233688